CLINICAL TRIAL: NCT05387993
Title: Incidence, Risk Factors and Microbiological Features of Infective Keratitis in Cairo University Hospitals
Brief Title: Microbial Keratitis in Cairo University Hospitals
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Nevien Lotfy Abdelkader, Ophthalmology Resident at the Ophthalmology Department, Cairo University., Kasr El Aini Hospital
Other Study IDs: MS-427-2020
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Infective Keratitis
Keywords: Corneal ulcer; Microbiological profile; Fungal keratitis; Bacterial keratitis; Infective keratitis; Antimicrobial susceptibility
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Corneal scrapings from cornea of infected eyes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to identify the incidence of infective keratitis presenting to the ophthalmology emergency department at Cairo University hospital, the risk factors and the bacterial/fungal spectrum causing the ulcers and to determine the best possible empirical therapy followed by specific therapy after obtaining culture results.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at the casualty who are clinically diagnosed as infectious keratitis , of all age groups and including both genders.

Exclusion Criteria:

Patients presenting with clinical picture suggestive of

* Viral keratitis solely without superimposed secondary infection.
* Non infectious keratitis as peripheral ulcerative keratitis ( e.g. Mooren's ulcer, marginal keratitis, autoimmune keratitis )

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment occurred from the Ophthalmology outpatient clinics and casualty department in Cairo University Hospitals, Kasr Al Aini.
  They met all inclusion and exclusion criteria for enrollment into this study.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
To identify risk factors and the most common causative organisms of microbial keratitis among the Egyptian population through history taking from each patient and the results of corneal sampling taken from the ulcer. | Three weeks for each participant
  Thorough history taking including risk factors that contributed to the ulcer occurrence. Corneal sampling through corneal scraping from the base and edge of the ulcer that undergoes direct examination and culturing using standard laboratory protocols.
To detect incidence of infective keratitis amongst all ophthalmological casualty cases by documenting the number of cases presenting or referred to the casualty of the ophthalmology department. | through study completion, an average of eight months
  Noting down the number of patients diagnosed with microbial keratitis that present to the casualty of a tertiary referral hospital, and calculate the percentage amongst all other ophthalmic casualty cases that present to the emergency as well.
To detect antimicrobial susceptibility and resistance of different antimicrobial agents causing corneal infections in our study group. | two weeks for each participant
  Antibiotic susceptibility testing was performed by the disc diffusion method (Modified Kirby Bauer technique) using Muller Hinton agar, aerobic incubation at 35°C for 16-18 hours. Anti fungal susceptibility was done using microdilution testing following the CLSI reference method.

SECONDARY OUTCOMES:
To assess the impact of culture and sensitivity results of corneal scrapings on the initial empirical therapy by calculating the number of cases that needed to shift the initial therapy to another one according to the antimicrobial susceptibility. | six months
  Empirical therapy according to the clinical impression that was shifted to another therapy according to the specific sensitivity results of positive growth cases.
Improving lines of management of microbial keratitis for a better outcome based on the cooperation between clinical ophthalmologists and microbiologists to reach a proper diagnosis and tailor the management accordingly. | six months
  Clinical impression of the nature of microbial keratitis , combined with the results of corneal scrapings positive growth cultures to detect the proper management plan for each patient to increase the chances of healed ulcers with medical therapy. Calculating the number of improving, healed and complicated cases.

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Mostafa, MD, Study Chair — Kasr Al Aini Hospital; Mohamed El Agha, MD, Study Director — Kasr Al Aini Hospital; Ihab Othman, MD, Study Director — Kasr Al Aini Hospital; Moushira Hosny, MD, Study Director — Kasr Al Aini Hospital; Nevien Lotfy, MSc, Principal Investigator — Kasr Al Aini Hospital
Locations (1):
- Kasr Al Aini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: After being published.